CLINICAL TRIAL: NCT06261502
Title: Effect of CANnabidiol on Anxiety and GABAergic Function in Individuals with Fragile-X Syndrome
Acronym: CANAX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Jazz Pharmaceuticals (Industry); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Francois Corbin, Full professor, Department of biochemistry, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-4527; 275882 (Other: Health Canada); 202010PJT-451514 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-01-26; First posted 2024-02-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Fragile X Syndrome
Keywords: FXS; CBD; TMS; MRI; eCB
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, placebo-controlled, single center, cross-over trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization and participant code allocation process will be carried out by the Centre de recherche du Centre hospitalier universitaire de Sherbrooke (CRCHUS) pharmacy. The pharmacy will dispense the medication or placebo based on the randomization. The principal investigators, Drs. Lepage and Corbin and the research, as well as the participants and their caregivers, will never be aware of the randomization. To avoid any suspicions on the part of the investigators, Dr. Artuela Çaku, who is not part of the research team, will have access to the laboratory results. In the event of an adverse drug effect, Dr. Çaku may break the code to make a more informed decision for the patient's well-being, such as discontinuing participation or reducing the dose, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBD First (Experimental): Participants will start with CBD to stimulate the eCB for 12 weeks, undergo an 8-week washout period, and then receive a 12-week placebo.
  Interventions: Drug: CBD Oral Solution; Drug: Placebo
- Placebo First (Experimental): Participants will start with a placebo for 12 weeks, undergo an 8-week washout period, and then receive a 12-week CBD to stimulate the eCB system.
  Interventions: Drug: CBD Oral Solution; Drug: Placebo

INTERVENTIONS:
Drug: CBD Oral Solution — Participants will start with oral CBD dose of 5 mg/kg/day for two weeks and then increase to 10 mg/kg/day.
Drug: Placebo — Participants will receive a dose of a placebo composed of the inactive ingredients of CBD of the same volume as the CBD Oral Solution.

SUMMARY:
This study focuses on the therapeutic relevance of the endocannabinoid (eCB) system for the treatment of Fragile-X syndrome (FXS), the primary hereditary cause of autism spectrum disorder (ASD). Most individuals with FXS have moderate to severe intellectual disability (ID), and caregivers are mainly concerned about aggressive behavior and anxiety problems. Since FXS individuals have a normal lifespan, the overall lifetime cost for the Canadian society of a single case is estimated at $1.2 to $4.7 millions reaching $18 billions for all FXS cases. There is no cure for FXS, as all clinical trials so far have been unsuccessful.FXS is caused by transcriptional silencing of the Fragile X mental retardation protein (FMR1) gene, making FXS a simple model to study ASD and ID pathophysiological mechanisms. Of those, neuronal hyperexcitability is largely recognized as a core deficit in FXS, and a critical therapeutic target for the disorder. Using transcranial magnetic stimulation (TMS) in FXS patients, our team provided the first direct evidence of Gamma-aminobutyric acid (GABA) receptor a (GABAa) dysfunctions in humans with this disorder and showed that this inhibitory deficit is linked with cortical hyperexcitability (PMID: 31748507). Concurrent lines of evidence suggest that stimulation of the endocannabinoid (eCB) system with the administration of Cannabidiol (CBD) could upregulate GABAergic function and correct inhibitory deficits presumed responsible for the neuropsychiatric phenotype of FXS. CBD has been shown to increase GABA concentration levels in the brains of healthy individuals, an effect that could help correct the hyperexcitability typically found in FXS. Thus, this trial aims to define the therapeutic potential of the eCB system for FXS, by measuring the impacts of oral CBD administration on the principal inhibitory neurotransmitter system of FXS patients, and the severity of the clinical phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of FXS
* Age 7 to 40 inclusively
* Overall ABC-C score > 20
* Taking up to 3 psychoactive drugs
* No therapeutic change for the last 3 months

Exclusion Criteria:

* Taking valproic acid
* Taking clobazam
* History of liver problems
* aspartate aminotransferase (AST) or alanine transaminase (ALT), > 3 times the reference values
* Bilirubin > 2 times the reference values
* Absolute contraindication to the use of TMS and MRI (e.g. presence of metal in the body), will also be considered as an exclusion criterion.

Ages: 7 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Oral CBD Solution anxiety. | At baseline, 12 weeks, 20 weeks, and 32 weeks
  Caregivers will complete The Anxiety, Depression, and Mood Scale (ADAMS). The ADAMS consists of 29 items on a 4-point scale from 0 (behavior have not occurred or is not a problem) to 3 (behavior occurs a lot, or is a severe problem). It evaluates emotional disturbances along five dimensions: mania/hyperactivity, depressed mood, social avoidance, general anxiety, and obsessive behavior.
Impact of Oral CBD Solution on disruptive behavior | At baseline, 12 weeks, 20 weeks, and 32 weeks
  Caregivers will complete the Aberrant Behavior Checklist-Community Fragile-X (ABC-C FX). The ABC-C FX has 55 items and is subdivided into explores 6 subdomains: irritability, hyperactivity, lethargy/withdrawal, stereotypy, inappropriate speech, and social avoidance. Higher scores reflect higher aberrant behavior.
  ABC-C FX is considered the gold standard for assessing behavioral changes in clinical trials in FXS.
Impact of Oral CBD Solution on Behavioral Inhibition | At baseline, 12 weeks, 20 weeks, and 32 weeks
  Participants will complete the NIH Toolbox Cognitive Battery Flanker Task, a behavioral inhibition task validated in FXS. Global scores range from 0 to 10 and are algorithmically defined using accuracy and reaction time. Higher scores reflect better performance.

SECONDARY OUTCOMES:
Impact of Oral CBD Solution on intracortical inhibition | At baseline, 12 weeks, 20 weeks, and 32 weeks
  TMS-derived measure of Intracortical inhibition: The degree of decrease of peak-to-peak motor evoked potential (MEP) amplitude induced by the administration of a conditioning stimulus (set at 70% of resting motor threshold) 2-4 ms before the test stimulus (stimulation intensity required to produce an MEP of 1 millivolt (mV), approximately 120% of resting motor threshold)
Impact of Oral CBD Solution on intracortical facilitation | At baseline, 12 weeks, 20 weeks, and 32 weeks
  Transcranial magnetic stimulation (TMS) -derived measure of Intracortical facilitation: The degree of increase of peak-to-peak motor evoked potential (MEP) amplitude induced by the administration of a conditioning stimulus (set at 80% of resting motor threshold) 12-24 ms before the test stimulus (stimulation intensity required to produce an MEP of 1 mV, approximately 120% of resting motor threshold).
Impact of Oral CBD Solution on | At baseline, 12 weeks, 20 weeks, and 32 weeks
  Estimation of GABA concentrations in the brain from magnetic resonance spectroscopy

IPD SHARING:
Plan to Share IPD: No